CLINICAL TRIAL: NCT02286245
Title: Effectiveness and Cost-effectiveness of Medical Advice Given by Telephone for Primary Care: the Formalised Telephone Medical Advice Study, a Cluster Randomised Control Trial.
Brief Title: The Effectiveness and Cost-effectiveness of Medical Advice Given by Telephone for Patients Calling for Primary Care
Acronym: CMTp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K120104; 2013-AO1722-43 (Other: IDRCB)
Record Dates: First submitted 2014-09-09; First posted 2014-11-07 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Isolated Fever; Gastroenteritis Symptoms
Keywords: Triage; Hotline; Primary Health Care; Emergency Medical Service Communication Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: focused Telephonic Medical Advice (Experimental): The physician will implement a protocol of care to each patient call for an isolated fever and/or symptoms of gastroenteritis: medical advice, drug prescription by phone and supervisory board. Patients are invited to recall in case of worsening or onset of new symptoms and to get an appointment with their general practitioner during working hours.
  Interventions: Other: focused Telephonic Medical Advice
- 2: Usual practice (Active Comparator): The physician will decide for the same disease (isolated fever and/or symptoms of gastroenteritis) the need of telephone advice with or without drug prescription, home visit by a doctor, emergency department services with or without EMS system.
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: focused Telephonic Medical Advice — The physician will implement a protocol of care to each patient call for an isolated fever and/or symptoms of gastroenteritis: medical advice, drug prescription by phone and supervisory board
  Arms: 1: focused Telephonic Medical Advice
Other: Usual practice — The physician will decide for the same disease (isolated fever and/or symptoms of gastroenteritis) the need of telephone advice with or without drug prescription, home visit by a doctor, emergency department services with or without EMS system.
  Arms: 2: Usual practice

SUMMARY:
Telephone medical advice in general practice is expanding. The Cochrane Database concludes in 2008 that there is not enough data about its use regarding out-of-hours general practitioners workload, emergency department visits, cost, safety and patient satisfaction. The aim of this study is to assess the effectiveness of telephone medical advice given by a general practitioner in a call centre for patient presenting isolated fever or gastroenteritis symptoms.

DETAILED DESCRIPTION:
This is a prospective, open label, cluster randomized trial of 2 880 expected patients who calling a French emergency medical service Dial 15 for fever or gastroenteritis symptoms during out-of-hours periods. All calls will be taken by a general practitioner (GP). Out-of-hours period is defined as 8 PM to 8 AM on weekdays, 1 PM to 8PM on Saturdays in addition to Sundays and holidays.To be exhaustive, we will enrol patients during one year.

In the experimental arm, the GP will implement a protocol of care to each patient call. The protocol includes medical advice, drug prescription by phone and supervisory board. Patients are invited to recall in case of worsening or onset of new symptoms and to get an appointment with their GP during working hours.

In the non-interventional arm, the GP will decide the need of telephone advice with or without drug prescription, home visit by a doctor, emergency department services with or without EMS system.

We will recall every patient at 15+/-4 days.

ELIGIBILITY:
Inclusion Criteria:

* Disease:

  * Fever: temperature ≥ 38 ° C
  * Symptoms of gastroenteritis include nausea and / or vomiting and / or diarrhea
* Onset of symptoms for less than 72 hours
* Age ≥ 18 years caller
* Patient age ≥ 1 year
* Affiliation to the French National Health Service

Exclusion Criteria:

* Pregnancy
* Severity criteria (fever> 41 ° C, disturbance of consciousness, rash, dyspnea, signs of dehydration, chest pain, neurological signs, gastrointestinal bleeding)
* Seeking advice from institutional correspondents (fire brigade, police, airport…)
* Communication difficulties (non-communicating patient, language barrier...)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2498 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patient with physical consultation by a general practitioner or in an emergency department, during out-of-hours periods | at 15 days
  Proportion of patient with physical consultation by a general practitioner or in an emergency department, during out-of-hours periods

SECONDARY OUTCOMES:
Cost effectiveness | at 15 days
  Cost effectiveness based on the economic analysis in each arm (sick leaves, hospitalization, EMS or firemen use...)
Care Mobile Units use | at 15 days
Emergency Medical Service use | at 15 days
Firemen use | at 15 days
  Number of fireman use
Recall at dispatching centre | at 15 days
Number and length of sick leave | at 15 days
All causes mortality | at 15 days
Morbidity | at 15 days
Patient satisfaction | at 15 days
  Patient satisfaction evaluated by a 14 items questionnaire ans a numeric scale from 0 to 10
Patient adhesion | at 15 days
  Percentage of patient's adhesion to the advice and/or drug prescriptions
Clinical outcome | at 15 days
  Percentage of relieved patients
Number of stay in intensive care unit | at 15 days
Number of hospitalisation | at 15 days
Number of patients seen repeatedly | at 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ADNET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SAMU 93 - EA 3409 - Faculté de Médecine de Bobigny - Université Paris 13, Bobigny, Île-de-France Region, France

REFERENCES:
- [Derived] Reuter PG, Durand-Zaleski I, Ducros O, Grignon O, Megy-Michoux I, Sourbes A, Desmettre T, Javaud N, Lapostolle F, Vicaut E, Adnet F. Efficacy of emergency medical center use of a protocol during telephone calls to give medical advice related to fever or gastroenteritis: a cluster randomized controlled trial. Emergencias. 2021 Aug;33(4):292-298. English, Spanish. PMID 34251142
- [Derived] Reuter PG, Desmettre T, Guinemer S, Ducros O, Begey S, Ricard-Hibon A, Billier L, Grignon O, Megy-Michoux I, Latouff JN, Sourbes A, Latier J, Durand-Zaleski I, Lapostolle F, Vicaut E, Adnet F. Effectiveness and cost-effectiveness of telephone consultations for fever or gastroenteritis using a formalised procedure in general practice: study protocol of a cluster randomised controlled trial. Trials. 2016 Sep 22;17(1):461. doi: 10.1186/s13063-016-1585-9. PMID 27659897